CLINICAL TRIAL: NCT00419926
Title: A Randomized, Multicenter, Parallel-group, Open-label Study to Evaluate the Therapeutic Benefit of an Initially Intensified Dosing Regimen of Mycophenolate Sodium Versus a Standard Dosing Regimen, in Combination With Cyclosporine and Corticosteroids in de Novo Renal Transplant Patients
Brief Title: Evaluation of the Therapeutic Benefit of an Initial Intensified Dosing Regimen of Mycophenolate Sodium Versus a Standard Regimen in Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2419
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Kidney Transplantation
Keywords: Renal, Kidney, Intensified, Enteric-coated mycophenolate sodium, Transplant
MeSH Terms: interventions — Mycophenolic Acid; Cyclosporine; Prednisone

ARMS (2):
- Intensified Mycophenolate Sodium (Myfortic) dosing regimen (Experimental): In patients randomized to the intensified Myfortic dosing regimen, the initial dose was 2-fold of the labeled dose (i.e. 2880 mg/day). The dosage was reduced to standard level in two steps,i.e. reduction to 2160 mg/day after 2 weeks of treatment and to 1440 mg/day after 6 weeks of treatment.
  Interventions: Drug: Enteric-coated mycophenolate sodium (Myfortic); Drug: Cyclosporine (Neoral); Drug: Prednisone
- Standard Mycophenolate Sodium (Myfortic) dosing regimen (Active Comparator): In patients randomized to the standard Myfortic dosing regimen, the initial dose of 1440 mg/day had to be maintained throughout the whole study.
  Interventions: Drug: Enteric-coated mycophenolate sodium (Myfortic); Drug: Cyclosporine (Neoral); Drug: Prednisone

INTERVENTIONS:
Drug: Enteric-coated mycophenolate sodium (Myfortic) — 1440 mg/day for the standard dose. 2880 mg/day for the initial intensified dosage, reduced to standard level in two steps,i.e. reduction to 2160 mg/day after 2 weeks of treatment and to 1440 mg/day after 6 weeks of treatment.
Drug: Cyclosporine (Neoral) — cyclosporine microemulsion in galenic form capsules starting at twice a day for a dose of 8-10 mg/kg/day adjusted if necessary to achieve protocol specific target levels
Drug: Prednisone — 20 mg orally per day reduced according to center practice for a minimum dose of 5 mg/day.

SUMMARY:
The purpose of this study is to determine if an initial intensified enteric-coated mycophenolate sodium (Myfortic) dosing regimen administered during the first six weeks post renal transplantation provides improved efficacy, with a similar safety profile, compared to a standard regimen of Myfortic.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 to 65 years old
* First or second time kidney transplant patients
* For females capable of becoming pregnant, negative pregnancy test prior to entry into trial and effective birth control during trial and 3 months after stopping trial medication

Exclusion Criteria:

* Previous graft loss due to immunological reasons in the 1st year after the 1st transplant
* Multi-organ recipients or previous transplant of another organ, different from the kidney
* Recipients from a non-heart-beating donor
* Known hypersensitivity to mycophenolic acid or cyclosporine
* HIV positive or Hepatitis B surface antigen positive
* History of malignancy (past 5 years)
* Pregnancy or planned pregnancy, lactating, or unwillingness to use effective contraception.
* Evidence of severe liver disease

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Mycophenolate Sodium (Myfortic) Dosing Regimen: In patients randomized to the standard Myfortic dosing regimen, the initial dose of 1440mg/day had to be maintained throughout the whole study.
Period: Overall Study
Arm/Group | Intensified Mycophenolate Sodium (Myfortic) Dosing Regimen | Standard Mycophenolate Sodium (Myfortic) Dosing Regimen
Started | 155 (Intention to treat population, 150 is safety population.) | 158 (Intention to treat population, 154 is safety population.)
Completed | 141 | 148
Not Completed | 14 | 10
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Administrative Problem | 4 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensified Mycophenolate Sodium (Myfortic) Dosing Regimen | Standard Mycophenolate Sodium (Myfortic) Dosing Regimen | Total
Number analyzed (Participants) | 155 | 158 | 313
Age, Customized [Number; unit: participants]
  < 50 years | 100 | 102 | 202
  >=50 years | 55 | 56 | 111
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 107
  Male | 102 | 104 | 206

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Failure 6-months Post Transplant Measured by the Combined Incidence of Biopsy Proven Acute Rejection, Graft Loss, and Death
Description: To evaluate therapeutic benefit by comparing the efficacy defined as the number of participants with treatment failure (biopsy-proven acute rejection [BPAR], graft loss [GFL] or death) at 6 months post-transplant. BPAR was defined as a biopsy graded IA, IB, IIA, IIB or III using Banff 2000 classification. A graft core biopsy was performed within 24 hours of initiation of anti-rejection therapy. GFL was defined as the day the allograft was presumed lost (the day the patient started dialysis, the day of nephrectomy or the day of irreversible graft loss demonstrated by imaging techniques.)
Time Frame: 6 months
Population: Intention to treat (ITT) population.
Measure: Number; unit: number of participants
Arm/Group | Intensified Mycophenolate Sodium (Myfortic) Dosing Regimen | Standard Mycophenolate Sodium (Myfortic) Dosing Regimen
Number analyzed (Participants) | 155 | 158
number of participants | 33 | 36

2. Secondary Outcome: Comparison of Overall Treatment Failure at Days 21 and 84 Post-transplantation Assessed by Biopsy Proven Acute Rejection (BPAR), GFL, and Death
Description: The overall treatment differences of the number of participants with at least one occurrence of the composite event BPAR, GFL or death at study days 21 and 84 post-transplantation. BPAR was defined as a biopsy graded IA, IB, IIA, IIB or III using Banff 2000 classification. A graft core biopsy was performed within 24 hours of initiation of anti-rejection therapy. GFL was defined as the day the allograft was presumed lost (the day the patient started dialysis, the day of nephrectomy or the day of irreversible graft loss demonstrated by imaging techniques.)
Time Frame: 21 and 84 days
Population: Intention to treat (ITT) population.
Measure: Number; unit: number of participants
Arm/Group | Intensified Mycophenolate Sodium (Myfortic) Dosing Regimen | Standard Mycophenolate Sodium (Myfortic) Dosing Regimen
Number analyzed (Participants) | 155 | 158
number of participants
  Day 21 | 20 | 21
  Day 84 | 33 | 34

3. Secondary Outcome: Comparison of Overall Treatment Failure at Days 21 and 84 Post-transplantation Assessed by Biopsy Proven Acute Rejection (BPAR), GFL, and Death
Description: as for outcome 2
Time Frame: 21 and 84 days
Population: Per Protocol (PP) population.
Measure: Number; unit: number of participants
Arm/Group | Intensified Mycophenolate Sodium (Myfortic) Dosing Regimen | Standard Mycophenolate Sodium (Myfortic) Dosing Regimen
Number analyzed (Participants) | 129 | 139
number of participants
  Day 21 | 14 | 20
  Day 84 | 26 | 33

4. Secondary Outcome: Renal Function Assessed by Glomerular Filtration Rate (GFR)at Each Visit
Description: The Modification of Diet in Renal Disease (MDRD) formula was used to calculate the GFR. Serum creatinine levels, age, sex and race were used to estimate the GFR levels in mL/min/1.73m^2.
Time Frame: at 21 days, 84 days and 180 days
Population: Intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: (mL/min/1.73m^2)
Arm/Group | Intensified Mycophenolate Sodium (Myfortic) Dosing Regimen | Standard Mycophenolate Sodium (Myfortic) Dosing Regimen
Number analyzed (Participants) | 155 | 158
(mL/min/1.73m^2)
  At 21 days | 47.3 (20.05) | 46.8 (21.00)
  At 84 days | 52.1 (19.80) | 51.8 (20.21)
  At 180 days | 53.5 (21.05) | 51.3 (25.14)

5. Secondary Outcome: Renal Function Assessed by Serum Creatinine at Each Visits
Time Frame: at 21 days, 84 days and 180 days
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: umol/L

6. Primary Outcome: Number of Patients With Treatment Failure 6-months Post Transplant Measured by the Combined Incidence of Biopsy Proven Acute Rejection, Graft Loss, and Death
Description: as for outcome 1
Time Frame: 6 months
Population: Per Protocol (PP) population.
Measure: Number; unit: number of participants
Arm/Group | Intensified Mycophenolate Sodium (Myfortic) Dosing Regimen | Standard Mycophenolate Sodium (Myfortic) Dosing Regimen
Number analyzed (Participants) | 129 | 139
number of participants | 26 | 35

ADVERSE EVENTS:
Arm/Group | Intensified Mycophenolate Sodium (Myfortic) Dosing Regimen | Standard Mycophenolate Sodium (Myfortic) Dosing Regimen
Serious Adverse Events (participants affected / at risk) | 74/150 | 68/154
Other Adverse Events (participants affected / at risk) | 143/150 | 145/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensified Mycophenolate Sodium (Myfortic) Dosing Regimen (N=150) | Standard Mycophenolate Sodium (Myfortic) Dosing Regimen (N=154)
Leukopenia (Blood and lymphatic system disorders) | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac hypertrophy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Kidney transplant rejection (Immune system disorders) | 1 | 7
Transplant rejection (Immune system disorders) | 0 | 1
BK virus infection (Infections and infestations) | 0 | 1
Cystitis escherichia (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 10 | 16
Cytomegalovirus syndrome (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Haematoma infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 2
Human polyomavirus infection (Infections and infestations) | 1 | 0
Incision site abscess (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 0 | 2
Infected lymphocele (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Renal cyst infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 9 | 11
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 6 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 2 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 | 2
Renal graft loss (Injury, poisoning and procedural complications) | 2 | 4
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 2 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound decomposition (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 5 | 5
Blood glucose increased (Investigations) | 0 | 1
Cytomegalovirus test (Investigations) | 1 | 0
Cytomegalovirus test positive (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Stupor (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Extravasation of urine (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 2
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 2 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urinary fistula (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urinoma (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 6
Lymphorrhoea (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intensified Mycophenolate Sodium (Myfortic) Dosing Regimen (N=150) | Standard Mycophenolate Sodium (Myfortic) Dosing Regimen (N=154)
Anaemia (Blood and lymphatic system disorders) | 39 | 37
Leukopenia (Blood and lymphatic system disorders) | 10 | 11
Tachycardia (Cardiac disorders) | 5 | 10
Abdominal discomfort (Gastrointestinal disorders) | 8 | 2
Abdominal distension (Gastrointestinal disorders) | 9 | 12
Abdominal pain (Gastrointestinal disorders) | 12 | 14
Abdominal pain upper (Gastrointestinal disorders) | 8 | 15
Constipation (Gastrointestinal disorders) | 58 | 51
Diarrhoea (Gastrointestinal disorders) | 40 | 27
Dyspepsia (Gastrointestinal disorders) | 10 | 7
Nausea (Gastrointestinal disorders) | 43 | 38
Vomiting (Gastrointestinal disorders) | 29 | 41
Fatigue (General disorders) | 8 | 3
Oedema (General disorders) | 5 | 12
Oedema peripheral (General disorders) | 42 | 46
Pain (General disorders) | 7 | 8
Pyrexia (General disorders) | 18 | 13
Kidney transplant rejection (Immune system disorders) | 4 | 8
Upper respiratory tract infection (Infections and infestations) | 15 | 11
Urinary tract infection (Infections and infestations) | 46 | 38
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 11 | 14
Incision site pain (Injury, poisoning and procedural complications) | 16 | 17
Procedural pain (Injury, poisoning and procedural complications) | 36 | 32
Blood creatinine increased (Investigations) | 14 | 20
Cytomegalovirus test positive (Investigations) | 9 | 4
Urine output decreased (Investigations) | 7 | 8
Weight increased (Investigations) | 1 | 8
Dehydration (Metabolism and nutrition disorders) | 8 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 12 | 12
Dyslipidaemia (Metabolism and nutrition disorders) | 8 | 10
Fluid overload (Metabolism and nutrition disorders) | 5 | 9
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 19
Hyperkalaemia (Metabolism and nutrition disorders) | 25 | 24
Hyperlipidaemia (Metabolism and nutrition disorders) | 14 | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 27
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 17 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 11
Dizziness (Nervous system disorders) | 9 | 7
Headache (Nervous system disorders) | 19 | 16
Paraesthesia (Nervous system disorders) | 6 | 11
Tremor (Nervous system disorders) | 19 | 20
Anxiety (Psychiatric disorders) | 8 | 12
Insomnia (Psychiatric disorders) | 21 | 23
Bladder spasm (Renal and urinary disorders) | 9 | 8
Dysuria (Renal and urinary disorders) | 17 | 13
Haematuria (Renal and urinary disorders) | 15 | 8
Renal tubular necrosis (Renal and urinary disorders) | 9 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 13
Acne (Skin and subcutaneous tissue disorders) | 9 | 9
Hirsutism (Skin and subcutaneous tissue disorders) | 8 | 6
Hypertrichosis (Skin and subcutaneous tissue disorders) | 3 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 9
Hypertension (Vascular disorders) | 51 | 45
Hypotension (Vascular disorders) | 11 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.